CLINICAL TRIAL: NCT07292311
Title: Reliability of Muscle Strength and Activation Assessment Tools and Effects of an Online Therapeutic Exercise Program in Patients With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Investigator, University of Extremadura
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 071125
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease; Renal Insufficiency, Chronic; Muscle Weakness; Sarcopenia; Physical Fitness; Physical Therapy Modalities
Keywords: chronic kidney disease; renal patients; muscle strength assessment; isokinetic testing; surface electromyography; physiotherapy; occupational therapy; functional evaluation; therapeutic exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Muscle Weakness; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reliability Assessment (Active Comparator): Test-retest reliability of isokinetic and surface EMG measurements in upper limb, trunk, and lower limb
  Interventions: Device: Reliability Assessment
- Online Therapeutic Exercise (Experimental): 8-10 week supervised online program including resistance and mobility exercises
  Interventions: Behavioral: Online Therapeutic Exercise

INTERVENTIONS:
Device: Reliability Assessment — Device: Isokinetic dynamometer and mDurance® surface EMG Test-retest reliability of isokinetic and surface EMG measurements in upper limb, trunk, and lower limb
  Arms: Reliability Assessment
Behavioral: Online Therapeutic Exercise — Behavioral: Online therapeutic exercise program 8-10 week supervised online program including resistance and mobility exercises
  Arms: Online Therapeutic Exercise

SUMMARY:
This research aims to evaluate the reliability and reproducibility of muscle strength and activation measurement tools, including isokinetic dynamometry and surface electromyography, in patients with chronic kidney disease (CKD). Additionally, the study will assess the feasibility and potential benefits of an online therapeutic exercise program supervised by physiotherapists.

DETAILED DESCRIPTION:
Patients with chronic kidney disease experience progressive muscle weakness and reduced physical capacity due to systemic inflammation, metabolic acidosis, and inactivity.

This two-phase observational and interventional study, conducted in collaboration with the ALCER Association (Badajoz and Cáceres, Spain), will:

1. Determine the test-retest reliability of muscle assessment tools (isokinetic dynamometer, surface electromyography, and handheld dynamometry).
2. Implement and evaluate an online therapeutic exercise program supervised by physiotherapists.

The project aims to provide valid and reliable protocols for neuromuscular assessment in CKD patients and explore the feasibility of remote therapeutic exercise.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Diagnosis of chronic kidney disease (hemodialysis, peritoneal dialysis, or kidney transplant).
* Member of ALCER Association (Badajoz or Cáceres).
* Medical clearance for physical testing/exercise.

Exclusion Criteria:

* Severe cognitive or communication impairment.
* Unstable cardiovascular or musculoskeletal conditions.
* Refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Test-retest reliability of surface EMG (Electromiography) activation. | 7-10 days
  RMS (root mean square). microvolts
Test-retest reliability of isokinetic strength | 7-10 days
  Intraclass Correlation Coefficient - ICC. Strength (kilograms)
Change in handgrip and limb strength measured by VALD dynamometry | Baseline and 12 weeks
  strength (kilograms)

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Enfermería y Terapia Ocupacional, Cáceres, Cáceres, Spain